CLINICAL TRIAL: NCT00285064
Title: Non-Invasive Assessment of Myocardial Viability Using Multidetector Computed Tomography Post Acute Myocardial Infarction
Brief Title: Assessment of Myocardial Viability Using Multidetector Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Philips Medical Systems (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ram1099_CTIL
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2007-02

CONDITIONS: Myocardial Infarction
Keywords: MDCT; viability
MeSH Terms: conditions — Myocardial Infarction

INTERVENTIONS:
Procedure: CT

SUMMARY:
To perform a comprehensive evaluation of multidetector CT myocardial enhancement patterns in patients with an acute ST elevation MI. In particular we plan to assess the relationship between regions with early hypoperfusion and/or late hyperenhancement, and myocardial viability.

DETAILED DESCRIPTION:
20 patients admitted to ICCU with ST elevation MI, and treated with primary angioplasty on admission, will undergo between day 2 and 7 post-MI the following exams: a) multidetector CT: regular scan plus late scan at 10 minutes, to evaluate coronary arteries, regional function and myocardial enhancement, b) echocardiography with echo-contrast to evaluate function and size of abnormally contracting region and remodeling, c) nuclear studies: rest early and late Thallium SPECT, to evaluate perfusion and viability. At 3 months a second echo will be performed to assess recovery of abnormal segments. The perfusion defects on MSCT will be compared with the other modalities and at 3 months will be used to evaluate recovery of myocardial function i.e. viability. Parameters that will be evaluated include opacity of hypoenhanced segments, ratio of normal to abnormal segments, change in opacity between early and late scans, size and transmurality of hypoenhanced segments, and their relation to regional contraction.

ELIGIBILITY:
Inclusion Criteria:

* acute ST elevation myocardial infarction
* after primary angioplasty

Exclusion Criteria:

* iodine allergy
* renal failure
* old MI
* arrhythmia
* inability to perform 20 second breath-hold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Prediction of viability from myocardial enhancement patterns

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lessick, MD DSc, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel